CLINICAL TRIAL: NCT02806076
Title: Radiofrequency Ablation Using Dual Cooled-Wet Electrode for Small Hepatocellular Carcinoma With No-touch Technique: Preliminary Study
Brief Title: RFA for Small HCC With No-touch Technique and Dual Cooled-Wet Electrode
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUH-2016-2243
Record Dates: First submitted 2016-06-03; First posted 2016-06-20 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No-touch RFA arm (Experimental): No-touch RFA arm indicates RFA procedure without direct tumor puncture. In this study, RFA is done by using dual cooled electrode.
  Interventions: Procedure: No-touch RFA arm
- Conventional tumor puncture RFA arm (Active Comparator): Conventional tumor puncture RFA arm indicates RFA procedure using "conventional tumor puncture" technique. In this study, RFA is done by using dual cooled electrode.
  Interventions: Procedure: Conventional tumor puncture RFA arm

INTERVENTIONS:
Procedure: No-touch RFA arm — No-touch RFA arm indicates RFA procedure without direct tumor puncture. In this study, RFA is done by using dual cooled electrode.
  Arms: No-touch RFA arm
Procedure: Conventional tumor puncture RFA arm — Conventional tumor puncture RFA arm indicates RFA procedure using "conventional tumor puncture" technique. In this study, RFA is done by using dual cooled electrode.
  Arms: Conventional tumor puncture RFA arm

SUMMARY:
The purpose of this study is to prospectively compare the clinical outcomes (local tumor progression rate, technical success rate, complication rate) of no touch radiofrequency ablation (RFA) technique for Hepatocellular carcinoma (HCC) to those of conventional tumor puncture RFA technique.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh class A
* patient with 1-2.5cm sized HCC
* 1 or 2 HCC lesions

Exclusion Criteria:

* maximum tumor diameter greater than 2.5cm
* Child-Pugh class B or C
* more than 3 HCC lesions
* invisible tumor even after US/CT or US/MR fusion
* presence of vascular tumor thrombosis or extrahepatic metastasis
* severe coagulopathy (PLT < 50K, PT < 50% of normal range)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
12 month local tumor progression (LTP) rate | 12 months after RFA

SECONDARY OUTCOMES:
2. tumor seeding rate | 12 months after RFA
Complication rate related with RFA | 1 month after RFA
  RFA-related complication rate such as death, abscess, bleeding..etc.
Technical success rate | 1 month after RFA
  presence or absence of residual lesion on follow-up imaging

OTHER OUTCOMES:
Ablation time | 3 days after RFA
  ablation time for tumor ablation
Intrahepatic distant mets | 12 months after RFA
  incidence of intrahepatic distant metastasis after RFA
Extrahepatic distant mets | 12 months after RFA
  incidence of extrahepatic distant metastasis after RFA
Technical efficacy 1 | 2 days after RFA
  Assessment of ablative margin using score 1-4 (1: residual tumor; 4: equal to or larger than 5mm) in side-by-side comparison of pre-RFA CT/MR and post-RFA CT using visual assessment
Technical efficacy 2 | 2 days after RFA
  Assessment of ablative margin using score 1-4 (1: residual tumor; 4: equal to or larger than 5mm) in side-by-side comparison of pre-RFA CT/MR and post-RFA CT using registration software

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No